CLINICAL TRIAL: NCT04126122
Title: Maternal and Neonatal Outcome in Severe Preeclamptic Patients
Brief Title: Maternal and Neonatal Outcome in Severe Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher , lecturer ,Obstetrics and Gynecology , National Research Centre, Aljazeera Hospital
Other Study IDs: Preeclampsia
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography to assess fetus and mother — to assess fetal growth and maternal outcome

SUMMARY:
In normal pregnancy the spiral arteries in the placental bed are invaded by trophoblast, which becomes incorporated into the vessel wall and replaces the endothelium, muscular layer and neural tissue

DETAILED DESCRIPTION:
Preeclampsia is considered severe if one or more of the following:

1. Blood pressure of 160mmHg systolic or high or 110mmHg diastolic or high on two occasions at least 6 hours a part while the patient on bed rest.
2. Proteinuria of 0.3gm. or high in 24 hours urine specimen or +1 or great on two random urine samples collected at least 4 hours apart.
3. Oliguria of less than 500ml in 24 hours.
4. Cerebral or visual disturbance.
5. Pulmonary edema or cyanosis.

ELIGIBILITY:
Inclusion Criteria:

* • All women with severe preeclampsia

Exclusion Criteria:

* • History of epilepsy.

  * Patients with chronic hypertension.
  * Patients with renal disease.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women with preeclampsia
Study Population: pregnant ladies with preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-01-10 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
The number of women who will develop adverse outcome | within 5 months
  The women with preeclampsia who will develop eclampsia or pulmonaryb edema

CONTACTS AND LOCATIONS:
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt